CLINICAL TRIAL: NCT00862186
Title: Self-Management of Cancer-Related Fatigue by Adolescents: Pilot Study of an Evidence Based Educational Resource
Brief Title: Self-Management of Cancer-Related Fatigue by Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Alex's Lemonade Stand Foundation (Industry)
Responsible Party: Principal Investigator, Catherine Fiona Macpherson, Investigator, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SCH-12551
Record Dates: First submitted 2009-03-12; First posted 2009-03-16 (Estimated); Results first posted 2012-05-09 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Neoplasms; Fatigue
Keywords: Neoplasms; Fatigue; Self Care
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Self-Management Arm (Other): Behavioral: 'Fatigue Facts & Fixes'
  Interventions: Behavioral: 'Fatigue Facts & Fixes'

INTERVENTIONS:
Behavioral: 'Fatigue Facts & Fixes' — 'Fatigue Facts & Fixes' is an evidence based educational resource for adolescents with cancer. It is a bright colored laminated 8.5x11 double sided page. One side features information on cancer-related fatigue: "Why am I so tired?" (description of cancer-related fatigue); "What causes fatigue?" (contributing factors - environmental, personal/behavioral, cultural/family/other, and treatment-related); and "What can help me to not be so tired?" (alleviating factors - environmental, personal/behavioral, cultural/family/other, and treatment-related). The other side is a 'Do Not Disturb' sign with a pillow graphic which adolescents can use in the hospital or at home when they need some quiet time and which may also serve to attract their interest to the resource.

SUMMARY:
This study will investigate self-management of cancer-related fatigue by adolescents through pilot study of an evidence based educational resource.

DETAILED DESCRIPTION:
Cancer-related fatigue is a prevalent and distressing symptom which has a significant impact on quality of life for children and adolescents with cancer and their families. Evidence based guidelines issued by the Oncology Nursing Society and National Comprehensive Cancer Network recommend educational interventions for preventing and treating cancer-related fatigue.The primary study aim is to examine the relationships among: intensity of cancer-related fatigue; frequency of use of an evidence based educational resource for self-management of cancer-related fatigue; and perceived helpfulness of resource use. The secondary aim is to examine the relationship between the Fatigue Scale-Adolescent (FS-A) and the Symptom Distress Scale (SDS) 'tired' item as measures of intensity of cancer-related fatigue. The tertiary aim is to examine the feasibility of recruiting and retaining adolescents with cancer for longitudinal study of cancer-related fatigue.

ELIGIBILITY:
Inclusion Criteria:

* adolescents 13-18 years inclusive
* leukemia, lymphoma, or malignant solid tumor; newly diagnosed and within 2 weeks of initiating therapy
* patient and consenting parent able to speak, read, and write English.

Exclusion Criteria:

* failure to meet all of inclusion criteria

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Fiona Macpherson, PhD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: 'Fatigue Facts & Fixes' is an evidence based educational resource for adolescents with cancer. It is a bright colored laminated 8.5x11 double sided page. One side features information on cancer-related fatigue: "Why am I so tired?" (description of cancer-related fatigue); "What causes fatigue?" (contributing factors - environmental, personal/behavioral, cultural/family/other, and treatment-related); and "What can help me to not be so tired?" (alleviating factors - environmental, personal/behavioral, cultural/family/other, and treatment-related). The other side is a 'Do Not Disturb' sign with a pillow graphic which adolescents can use in the hospital or at home when they need some quiet time and which may also serve to attract their interest to the resource.
Period: Overall Study
Arm/Group | Group 1
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 13.33 (3.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fatigue Scale-Adolescent (FS-A) Score Categorized According to 1-5 Rating Scale of Resource Use and Resource Helpfulness.
Description: The FS-A is a 14-item self-report instrument which measures on a 5 point scale ranging from '1 - not at all' to '5 - all the time' the extent to which each of 14 statements describes how the respondent has been feeling during the past 7 days (Hinds et al., 2007). The potential score range is 14-70; higher scores represent greater fatigue (Hinds et al., 2007). The scores (1 through 5) on the Likert-type scales for resource use and resource helpfulness were determined at each post baseline time point, as were change from baseline values for the FS-A. All FS-A change from baseline values, per Resource Use or Resource Helpfulness Categorization, were combined regardless of post-baseline time point.
Time Frame: baseline and weekly up to 8 weeks
Measure: Median (Full Range); unit: units on a scale
Groups:
- Resource Use: Fatigue Facts & Fixes was assessed for amount of resource use on a 1-5 Likert-type scale.
- Resource Helpfulness: Fatigue Facts & Fixes was assessed for amount of resource helpfulness on a 1-5 Likert-type scale.
Arm/Group | Resource Use | Resource Helpfulness
Number analyzed (Participants) | 15 | 15
units on a scale
  1 - not at all | -3 [-32 to 10] | -3 [-32 to 10]
  2 - | -4 [-24 to 2] | -4 [-24 to 1]
  3- | -4 [-19 to 10] | -7 [-30 to 9]
  4 - | -8.5 [-31 to -3] | -2.5 [-31 to 10]
  5 - a lot | -1 [-13 to 0] | -4 [-17 to 0]

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
Slow enrollment resulting in low accrual - only 15 participants rather than the 60 planned - therefore unable to complete analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes